CLINICAL TRIAL: NCT02446444
Title: Randomised Phase 3 Trial of Enzalutamide in Androgen Deprivation Therapy With Radiation Therapy for High Risk, Clinically Localised, Prostate Cancer: ENZARAD
Brief Title: Enzalutamide in Androgen Deprivation Therapy With Radiation Therapy for High Risk, Clinically Localised, Prostate Cancer
Acronym: ENZARAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); National Health and Medical Research Council, Australia (Other); Cancer Trials Ireland (Network); Trans Tasman Radiation Oncology Group (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANZUP1303; ACTRN12614000126617 (Other: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2015-05-04; First posted 2015-05-18 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms
Keywords: High risk; clinically localised prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Stratification Factors:
  * Gleason score (<=7 versus 8-10),
  * Regional lymph nodes involvement (N0 versus N1)
  * Clinical T-stage (T2 and below versus T3 and above),
  * PSA (<20ng/mL versus ≥ 20ng/mL)
  * Study Site
  * Brachytherapy (yes versus no)
  * Pelvic Field (yes versus no)
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enzalutamide (Experimental): Enzalutamide 160 mg daily, by mouth, for 24 months from randomisation. All participants are treated with a LHRHA for 24 months from randomisation and external beam radiation therapy started approximately 16 weeks after randomisation (+/- brachytherapy boost)
  Interventions: Drug: Enzalutamide; Drug: LHRHA; Radiation: External Beam Radiotherapy (78 Gy in 39 fractions or 46 Gy in 23 fractions plus brachytherapy boost)
- Conventional Non-steroidal Anti-androgen (NSAA) (Active Comparator): Conventional Non-steroidal Anti-androgen (NSAA), by mouth, for 6 months from randomisation.
  All participants are treated with a LHRHA for 24 months from randomisation and external beam radiation therapy started approximately 16 weeks after randomisation (+/- brachytherapy boost)
  Interventions: Drug: Conventional NSAA; Drug: LHRHA; Radiation: External Beam Radiotherapy (78 Gy in 39 fractions or 46 Gy in 23 fractions plus brachytherapy boost)

INTERVENTIONS:
Drug: Enzalutamide
  Arms: Enzalutamide
Drug: Conventional NSAA
  Arms: Conventional Non-steroidal Anti-androgen (NSAA)
Drug: LHRHA
Radiation: External Beam Radiotherapy (78 Gy in 39 fractions or 46 Gy in 23 fractions plus brachytherapy boost)

SUMMARY:
The purpose of this study is to determine the effectiveness of enzalutamide as part of adjuvant androgen deprivation therapy (ADT) with a luteinizing hormone releasing hormone analogue (LHRHA) in men having radiation therapy for localised prostate cancer at high risk of recurrence.

ELIGIBILITY:
Men with localised prostate cancer at high risk for recurrence deemed suitable for external beam radiation therapy.

Inclusion Criteria:

1. Pathological diagnosis of adenocarcinoma of the prostate, judged to be at high risk for recurrence based on any of the following (in accordance with the International Society of Urological Pathology (ISUP) Consensus 2005:

   Gleason score 8-10 OR Gleason score of 4+3 AND clinical T2b-4 AND PSA >20ng/mL OR N1 disease (involvement of lymph nodes at or below the bifurcation of the common iliac arteries) defined radiologically as greater than 10mm on short axis using standard CT or MRI, or biopsy proven
2. Age ≥18 years
3. Adequate bone marrow function Haemoglobin (Hb) ≥100g/L and White Cell Count (WCC) ≥ 4.0 x 109/L and platelets ≥100 x 109/L
4. Adequate liver function: Alanine transaminase (ALT) < 2 x ULN and bilirubin < 1.5 x Upper Limit of Normal (ULN), (or if bilirubin is between 1.5 - 2 x ULN, they must have a normal conjugated bilirubin).
5. Adequate renal function: calculated creatinine clearance > 30 ml/min (Cockcroft-Gault)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
7. Study treatment both planned and able to start within 7 days of randomisation.
8. Willing and able to comply with all study requirements, including treatment, and attending required assessments
9. Has completed the baseline HRQOL questionnaires UNLESS is unable to complete because of literacy or limited vision
10. Signed, written, informed consent

Exclusion Criteria:

1. Prostate cancer with significant sarcomatoid or spindle cell or neuroendocrine small cell components
2. Involvement of lymph nodes superior to the common iliac bifurcation, and/or outside the pelvis (distant lymph nodes). Lymph node involvement is defined by histopathological confirmation, or by a short axis measurement >10mm on standard imaging (CT or MRI, but not PET).
3. Any contraindication to external beam radiotherapy
4. History of

   * seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma).
   * loss of consciousness or transient ischemic attack within 12 months of randomization
   * significant cardiovascular disease within the last 3 months: including myocardial infarction, unstable angina, congestive heart failure (NYHA grade II or greater), ongoing arrhythmias of Grade > 2 , thromboembolic events (e.g., deep vein thrombosis, pulmonary embolism). Chronic stable atrial fibrillation on stable anticoagulant therapy is allowed.
5. Evidence of metastatic disease: minimum imaging required Computed tomography scan (CT) / Magnetic Resonance Imaging (MRI) of the abdomen and pelvis, and Whole Body Bone Scan (WBBS). If equivocal bone scan, follow-up plain films are required to show NO evidence of cancer if not covered by CT/MRI
6. PSA > 100 ng/mL
7. History of another malignancy within 5 years prior to randomisation except for non-melanomatous carcinoma of the skin; or, adequately treated, non-muscle-invasive urothelial carcinoma of the bladder (i.e. Tis, Ta and low grade T1 tumours).
8. Concurrent illness, including severe infection that might jeopardize the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety

   * Human Immunodeficiency Virus (HIV)-infection is not an exclusion criterion if it is controlled with anti-retroviral drugs that are unaffected by concomitant enzalutamide.
9. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule, including alcohol dependence or drug abuse;
10. Patients who are sexually active and not willing/able to use medically acceptable forms of barrier contraception.
11. Use of hormonal therapy or androgen deprivation therapy, including enzalutamide, except in the following setting:

    * Use of LHRHA (with or without anti-androgens) for less than 30 days prior to randomisation in the trial.
12. Bilateral orchidectomy or radical prostatectomy
13. Prior brachytherapy or other radiotherapy that would result in an overlap of radiotherapy fields
14. Participation in other clinical trials of investigational agents for the treatment of prostate cancer or other diseases.
15. Major surgery within 21 days prior to randomisation
16. Known gastrointestinal (GI) disease or GI procedure that could interfere with the oral absorption or tolerance of enzalutamide, including difficulty swallowing tablets

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2014-03; Primary Completion 2025-06 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Metastasis-free survival | 5 years
  Metastasis free survival (MFS) is defined as the interval from the date of randomisation to the date of first evidence of metastasis or death from any cause, whichever occurs first, or the date of last known follow-up alive and without metastases.
  Evidence of metastasis includes findings on whole body bone scan (WBBS) or CT or MRI that are either characteristic of metastatic prostate cancer, and/or confirmed by other test results, e.g. cytology or histopathology, and lesion qualifies as new metastatic disease per RECIST 1.1. Detection of metastasis by other modalities, eg Ga-68 PSMA (Prostate Specific Membrane Antigen) PET, does not constitute an event unless confirmed by WBBS or CT or MR

SECONDARY OUTCOMES:
Overall survival | 5 years
  Overall survival (OS) is defined as the interval from the date of randomisation to date of death from any cause, or the date of last known follow-up alive.
Prostate cancer-specific survival | 5 years
  Prostate cancer-specific survival is defined as the interval from the date of randomisation to the date of death from prostate cancer, or the date of last known follow-up alive.
PSA (Prostate-Specific Antigen) progression-free survival | 5 years
  PSA progression-free survival is defined as the interval from the date of randomisation to the date of first evidence of PSA progression, clinical progression, or death from any cause, whichever occurs first, or the date of last known follow-up without PSA progression and without clinical progression.
  PSA progression as defined by the Phoenix criteria: an increase in PSA of more than 2ng/mL above the nadir (lowest) PSA level.
Clinical progression-free survival | 5 years
  Clinical progression-free survival is defined as the interval from the date of randomisation to the date of first clinical evidence of disease progression or death from any cause, whichever occurs first, or the date of last known follow-up alive without clinical progression.
  Clinical evidence of disease progression includes evidence of progression or recurrence on imaging, clinical examination, development of symptoms attributable to cancer progression, or initiation of other anticancer treatment for prostate cancer.
Time to subsequent hormonal therapy | 5 years
  Time to subsequent hormone therapy is the interval from randomisation to the first date that androgen deprivation therapy is recommenced for the treatment of recurrent (or progressive) prostate cancer, or the date of last known follow-up without recommencement of androgen deprivation therapy.
Time to castration-resistant disease (PCWG2 criteria) | 5 years
  Castration resistant prostate cancer (CRPC) is defined, per PCWG2, by a rising PSA that is greater than 2ng/mL higher than the most recent nadir with a testosterone < 50 ng/dL (<1.7 nmol/L); the rise has to be at least 25% over the most recent nadir; and, the rise has to be confirmed by a second PSA at least three weeks later. The time to castration-resistant prostate cancer is defined as the interval from randomisation to the date that the PSA first met the criteria defined above (i.e. the date of the first PSA to meet these criteria, not the date of the subsequent confirmatory test), or the date of last known follow-up without CRPC.
Safety (adverse events - CTCAE v4.03) | 5 years
  The NCI Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE v4.03) will be used to classify and grade the intensity of adverse events occurring until 30 days after the last dose of study treatment.
Health related quality of life (HRQL) | 5 years
  HRQL will be reported by participants using the EORTC core quality of life questionnaire (QLQ C-30) and prostate cancer specific module (PR-25). The EQ-5D-5L will be used to derive utility scores suitable for quality adjusted survival analyses
Health outcomes relative to costs (incremental cost effectiveness ratio) | 5 years
  Information on the following areas of health-care resource usage will be collected: hospitalisations, visits to health professionals, and medications. Quality-adjusted survival (QAS) time will be used to quantify the incremental effectiveness of adding enzalutamide to standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Williams, Study Chair — ANZUP and Peter MacCallum Cancer Centre; Paul Nguyen, Study Chair — Dana Farber Cancer Institute and ANZUP
Locations (69):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
- Australia (41):
  - Blacktown Hospital, Blacktown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Genesis Cancer Care Newcastle, Gateshead, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Tamworth Rural Referral Hospital, Tamworth, New South Wales
  - Sydney Adventist Hospital, Wahroonga, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Genesis Cancer Care Queensland - Wesley and Chermside, Auchenflower, Queensland
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane & Womens Hospital, Herston, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Radiation Oncology Services Mater Centre, South Brisbane, Queensland
  - ICON - Gold Coast (formerly ROC Gold Coast), Southport, Queensland
  - ICON - Toowoomba (formerly ROC Toowoomba), Toowoomba, Queensland
  - Genesis Cancer Care Queensland - Tugun and Southport, Tugun, Queensland
  - Princess Alexandra Hospital Brisbane, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research (Adelaide Cancer Centre), Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Peter MacCallum Cancer Centre, Bendigo, Victoria
  - Peter MacCallum Cancer Centre (Moorabbin Campus), Bentleigh East, Victoria
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
  - Genesis Care - Epping (formerly EROC), Epping, Victoria
  - Genesis Care - Western (formerly WROC), Footscray, Victoria
  - Genesis Care - Frankston (formerly FROC), Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Epworth HealthCare - Richmond, Richmond, Victoria
  - Genesis Care - Ringwood (formerly RROC), Ringwood East, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Salzburger Landeskliniken - Universitätsklinikum Salzburg, Salzburg, Austria
- AZ Groeninge Kortrijk- Campus Kennedylaan, Kortrijk, Belgium
- Ireland (6):
  - Cork University Hospital, Cork, Co Cork
  - Galway University Hospital, Galway, Co Galway
  - Mater Misericordiae University Hospital, Dublin, Dublin 7
  - Beacon Private Hospital, Dublin
  - St Luke's Hospital, Dublin
  - Mater Private Hospital, Dublin
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
- The Institute Of Oncology, Ljubljana, Slovenia
- Spain (3):
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Badalona, Barcelona
  - Hospital Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (11):
  - Velindre Hospital, Whitchurch, Cardiff
  - University Hospital Southhampton, Southampton, Hampshire
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Royal Marsden Hospital, Chelsea, London
  - Western General Hospital, Edinburgh, Scotland
  - Royal United Hospital Bath, Bath
  - Addenbrookes Hospital, Cambridge
  - University of London Hospital, London
  - Guys and St Thomas Hospital, London
  - Charring Cross Hospital: Imperial College Healthcare NHS Trust, London
  - Nottingham City Hospital- City Campus, Nottingham

REFERENCES:
- See also: Australian and New Zealand Urogenital and Prostate (ANZUP) Cancer Trials Group. — https://www.anzup.org.au
- See also: University of Sydney, National Health and Medical Research Council (NHMRC) Clinical Trials Centre. — http://ctc.usyd.edu.au/
- See also: Australian New Zealand Clinical Trials Registry (ANZCTR) — http://www.anzctr.org.au/